CLINICAL TRIAL: NCT06410469
Title: A Novel Suturing Technique for Natural Tissue Repair in Cystocele Treatment
Brief Title: A Novel Suturing Technique of Cystocele Treatment
Acronym: cystosel
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Rahime Bedir Fındık, Associate Professor Dr, Ankara City Hospital Bilkent
Other Study IDs: AnkaraCHBilkent-MH-RBF-04
Record Dates: First submitted 2024-05-03; First posted 2024-05-13 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Cystocele
Keywords: anterior colporraphy; naturel tissue; suture technique
MeSH Terms: conditions — Cystocele

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 33 patients operated with rug wave: Group1
  Interventions: Procedure: rug weaving-like plication technique
- 32 patients who underwent surgery using conventional colporrhaphy.: Group 2

INTERVENTIONS:
Procedure: rug weaving-like plication technique — anterior vaginal wall repair with the rug weaving-like plication technique in cystosel
  Groups: 33 patients operated with rug wave

SUMMARY:
The rug weaving-like plication technique may offer a viable alternative for cystocele repair without mesh, utilizing natural tissue.

DETAILED DESCRIPTION:
The aim of this study is to compare patients who underwent cystocele repair using the rug weaving plication technique, a natural tissue repair method implemented since 2022 for anterior prolapse, with those treated using conventional techniques.

The investigators retrospectively reviewed 33 patients who underwent anterior vaginal wall repair with the rug weaving-like plication technique and 32 patients who underwent surgery using conventional colporrhaphy. The investigators recorded demographic data and operative details of the patients. At the 6-month postoperative follow-up,the investigators assessed patients' complaints, Pelvic Organ Prolapse Quantification (POP-Q), Modified Oxford Scoring (MOS), and pelvic floor muscle strength. The investigators measured bladder wall thickness between the bladder and anterior vaginal wall using Transvaginal Ultrasonography (USG) and compared demographic data, operative details, and postoperative outcomes between the two groups.

ELIGIBILITY:
Inclusion Criteria: Patients operated on using the rug weaving plication technique

Exclusion Criteria:Patients operated on using the conventional anterior colporrhaphy

Ages: 40 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Results of cystocele surgery in women
Study Population: Women operated on for anterior wall prolapse in POP-Q
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Quantification (POP-Q) | Maximum 6 months
  Postoperative anterior wall POP-Q
  Measurements were conducted with a scaled abeslang while the patient was in the lithotomy position. Evaluation of the anterior compartment involved measuring points Aa and Ba, the apical compartment involved points C and D, and the posterior compartment involved points Ap and Bp. Staging was determined based on the lowest point of prolapse. Stage 0 indicated normal pelvic floor support, Stage 2 indicated a distance between -1 and 1 from the hymen, and Stage 4 indicated total uterine prolapse (prosidentia). Stages 1,2 and 3 indicated intermediary levels of prolapse severity, counting for grades between Stage 0 and 4.

SECONDARY OUTCOMES:
Bladder thickness | Maximum 6 months
  Postoperative bladder thickness:Bladder wall thickness between the bladder and anterior vaginal wall was measured using transvaginal ultrasonography and recorded in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Rahime Bedir Findik, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Findik RB, Doganay M, Aksakal OS, Coskun ZY, Karakaya J. A novel suturing technique for natural tissue repair in cystocele treatment. BMC Womens Health. 2024 Aug 29;24(1):474. doi: 10.1186/s12905-024-03317-3. PMID 39210362